CLINICAL TRIAL: NCT01801436
Title: A Post Approval Commitment Study for Pharmacokinetic Analysis and Providing Expanded Access to Bortezomib (Velcade) for Patients With Multiple Myeloma Who Have Received at Least Two Previous Lines of Therapy and Are Refractory to or Have Relapsed After Their Last Therapy for Multiple Myeloma in Taiwan
Brief Title: A Post-Approval Pharmacokinetic Study of Bortezomib in Participants With Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Taiwan Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013843; 26866138MMY3014
Record Dates: First submitted 2013-02-27; First posted 2013-02-28 (Estimated); Results first posted 2013-05-16 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-03

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Bortezomib; Velcade
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bortezomib (Experimental): Bortezomib 1.3 milligram (mg) per meter square (m^2) on Days 1, 4, 8, and 11 of each 3-week cycle for up to 8 cycles.
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Bortezomib 1.3 mg per (m^2) on Days 1, 4, 8, and 11 of each 3-week cycle for up to 8 cycles.
  Other Names: VELCADE

SUMMARY:
The purpose of this post marketing study is to determine the plasma concentration of bortezomib (unchanged drug) to assess the pharmacokinetic (PK - the study of the way a drug enters and leaves the blood and tissues over time) properties in the Taiwanese population. It will also provide expanded access (expanded access, sometimes called "compassionate use," is the use of an investigational drug outside of a clinical trial to treat a participant with a serious or immediately life-threatening disease or condition who has no comparable or satisfactory alternative treatment options) to bortezomib for the same group of participants with multiple myeloma (cancer of the types of cells normally found in bone marrow).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single-arm, multi-center (conducted in more than 1 center) study to assess the PK of bortezomib and to provide expanded access to bortezomib for 14 Taiwanese participants with multiple myeloma who have received at least 2 previous lines of therapy (medicine or medical care given to a participant for a disease or condition) and are refractory (not responding to treatment) to or have relapsed (the return of a medical problem) after their last therapy. Eligible participants will receive bortezomib 1.3 milligram (mg) per meter square (m^2) on Days 1, 4, 8, and 11 of each 3-week cycle for up to 8 cycles. Blood samples for PK assessment will be collected on specified time points of Day 1, Day 8, and Day 11 of Cycle 1. Efficacy of the participants will primarily be evaluated by recording 'response to treatment' and 'Karnofsky Performance Status'. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants previously diagnosed with multiple myeloma based on standard criteria
* Participant has received at least 2 previous lines of therapy for multiple myeloma and, in the Investigator's opinion, currently requires therapy because of relapsed (the return of a medical problem) or progressive disease
* Female participants either postmenopausal or surgically sterilized or willing to use an acceptable method of birth control from Screening through the Final Visit
* If male, the participant agrees to use an acceptable barrier method for contraception from Screening through the Final Visit
* Participant has a Karnofsky performance status classifies participants as to their functional impairment and is used to compare effectiveness of different therapies and to assess the prognosis [outlook, probable outcomes] in individual participants) greater than 60

Exclusion Criteria:

* If the participant received bortezomib in a previous trial, the Participants' best response to bortezomib must be progressive disease
* If the participant received bortezomib in a previous trial, the participant must have experienced 1 or more serious adverse events
* Participants who have received nitrosoureas within 6 weeks or any other chemotherapy (treatment of disease, usually cancer, by chemical agents) within 3 weeks before enrollment
* Participants who have received corticosteroids (greater than 10 milligram per day prednisone or equivalent) within 3 weeks before enrollment
* Human Immunodeficiency Virus (HIV - a life-threatening infection which you can get from an infected person's blood or from having sex with an infected person)-positive or hepatitis-B surface antigen-positive participants or participants with known active hepatitis-C infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-12; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Taiwan Ltd Clinical Trial, Study Director — Johnson & Johnson Taiwan Ltd

RESULTS

PARTICIPANT FLOW:
Groups:
- Bortezomib: Participants received 1.3 milligram per meter square (mg per m^2) of bortezomib on Days 1, 4, 8, and 11 of each 3-week cycle for up to 8 cycles.
Period: Overall Study
Arm/Group | Bortezomib
Started | 14
Completed | 5
Not Completed | 9
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 2
Not completed — Progressive disease | 4

BASELINE CHARACTERISTICS:
Groups:
- Bortezomib: Participants received 1.3 mg per m^2 of bortezomib on Days 1, 4, 8, and 11 of each 3-week cycle for up to 8 cycles.
Arm/Group | Bortezomib
Number analyzed (Participants) | 14
Age Continuous [Mean (Standard Deviation); unit: Years] | 62.63 (8.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response to Treatment at Day 1 of Cycle 5
Description: Response to treatment was based on the changes in monoclonal protein (M-protein) in serum and urine. Response categories were complete response: complete clearance of M-protein for at least 6 weeks, response: at least 75 percent reduction in M-protein for at least 2 determinations 6 weeks apart, partial response: 50 to 74 percent reduction in M-protein, minimal response: 25 to 49 percent reduction in M-protein, stable disease: not qualifying minimal response or progression and progression: increased M-protein level in serum or urine or clinical signs of disease progression.
Time Frame: Day 1 of Cycle 5
Population: The full analysis set (FAS) population included all the participants who received 1 dose of study medication and had post-dose efficacy data. Here 'N' signifies those participants who were evaluated for this outcome measures.
Measure: Number; unit: Participants
Arm/Group | Bortezomib
Number analyzed (Participants) | 7
Participants
  Complete response | 1
  Response | 2
  Partial Response | 2
  Stable disease | 1
  Progression | 1

2. Primary Outcome: Number of Participants With Response to Treatment at Day 1 of Cycle 7
Description: as for outcome 1
Time Frame: Day 1 of Cycle 7
Population: The FAS population included all the participants who received 1 dose of study medication and had post-dose efficacy data. Here 'N' signifies those participants who were evaluated for this outcome measures.
Measure: Number; unit: Participants
Arm/Group | Bortezomib
Number analyzed (Participants) | 5
Participants
  Response | 1
  Partial Response | 3
  Stable disease | 1

3. Primary Outcome: Number of Participants With Response to Treatment at Day 11 of Cycle 8
Description: as for outcome 1
Time Frame: Day 11 of Cycle 8
Population: The FAS population included all the participants who received 1 dose of study medication and had post-dose efficacy data.
Measure: Number; unit: Participants
Arm/Group | Bortezomib
Number analyzed (Participants) | 14
Participants
  Response | 2
  Partial response | 3
  Minimal response | 2
  Stable disease | 1
  Progression | 6

4. Primary Outcome: Number of Participants With Karnofsky Performance Status (KPS) Score at Baseline
Description: The KPS Index allows participants to be classified as per their functional impairment (abnormal function). This can be used to compare effectiveness of different therapies (medicine or medical care given to a participant for a disease or condition) and to assess the prognosis (outlook, probable outcomes) in individual participants. KPS was recorded on an 11-point scale (0, 10, 20, 30, 40, 50, 60, 70, 80, 90, and 100.) where '0=Dead' and '100=Normal, no complaints, no evidence of disease'. The lower the Karnofsky score, the worse the survival for most serious illnesses.
Time Frame: Baseline
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Bortezomib
Number analyzed (Participants) | 14
Participants
  KPS Score = 70 | 2
  KPS Score = 80 | 3
  KPS Score = 90 | 7
  KPS Score = 100 | 2

5. Primary Outcome: Number of Participants With KPS Score at Day 1 of Cycle 1
Description: as for outcome 4
Time Frame: Day 1 of Cycle 1
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Bortezomib
Number analyzed (Participants) | 14
Participants
  KPS Score = 70 | 2
  KPS Score = 80 | 5
  KPS Score = 90 | 5
  KPS Score = 100 | 2

6. Primary Outcome: Number of Participants With KPS Score at Day 1 of Cycle 3
Description: as for outcome 4
Time Frame: Day 1 of Cycle 3
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Bortezomib
Number analyzed (Participants) | 12
Participants
  KPS Score = 60 | 1
  KPS Score = 70 | 1
  KPS Score = 80 | 6
  KPS Score = 90 | 2
  KPS Score = 100 | 2

7. Primary Outcome: Number of Participants With KPS Score at Day 1 of Cycle 5
Description: as for outcome 4
Time Frame: Day 1 of Cycle 5
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Bortezomib
Number analyzed (Participants) | 7
Participants
  KPS Score = 60 | 1
  KPS Score = 70 | 1
  KPS Score = 80 | 4
  KPS Score = 100 | 1

8. Primary Outcome: Number of Participants With KPS Score at Day 1 of Cycle 7
Description: as for outcome 4
Time Frame: Day 1 of Cycle 7
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Bortezomib
Number analyzed (Participants) | 5
Participants
  KPS Score = 60 | 1
  KPS Score = 80 | 2
  KPS Score = 90 | 1
  KPS Score = 100 | 1

9. Primary Outcome: Number of Participants With KPS Score at Day 11 of Cycle 8
Description: as for outcome 4
Time Frame: Day 11 of Cycle 8
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Bortezomib
Number analyzed (Participants) | 14
Participants
  KPS Score = 50 | 2
  KPS Score = 60 | 4
  KPS Score = 70 | 1
  KPS Score = 80 | 3
  KPS Score = 90 | 2
  KPS Score = 100 | 2

10. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Bortezomib on Day 1 of Cycle 1
Description: The Cmax is observed maximum plasma concentration, taken directly from the plasma concentration-time profile.
Time Frame: 0 hour (Pre-dose) and 0.08, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours (post-dose) on Day 1 of Cycle 1
Population: The Per-protocol (PP) population included all the participants who received study medications as per the administration schedule and for whom blood samples were collected at all scheduled time points.
Measure: Mean (Standard Deviation); unit: Nanogram per millileter (ng per ml)
Arm/Group | Bortezomib
Number analyzed (Participants) | 10
Nanogram per millileter (ng per ml) | 76.43 (38.47)

11. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Bortezomib on Day 11 of Cycle 1
Description: The Cmax is observed maximum plasma concentration, taken directly from the plasma concentration-time profile.
Time Frame: 0 hour (Pre-dose) and 0.08, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours (post-dose) on Day 11 of Cycle 1
Population: The PP population included all the participants who received study medications as per the administration schedule and for whom blood samples were collected at all scheduled time points.
Measure: Mean (Standard Deviation); unit: ng per ml
Arm/Group | Bortezomib
Number analyzed (Participants) | 10
ng per ml | 127.02 (59.80)

12. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Bortezomib on Day 1 of Cycle 1
Description: Tmax is the time when Cmax is observed, taken directly from the plasma concentration-time profile.
Time Frame: 0 hour (Pre-dose) and 0.08, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours (post-dose) on Day 1 of Cycle 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Bortezomib
Number analyzed (Participants) | 10
Hours | 0.08 (0.00)

13. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Bortezomib on Day 11 of Cycle 1
Description: Tmax is the time when Cmax is observed, taken directly from the plasma concentration-time profile.
Time Frame: 0 hour (Pre-dose) and 0.08, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours (post-dose) on Day 11 of Cycle 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Bortezomib
Number analyzed (Participants) | 10
Hours | 0.08 (0.01)

14. Primary Outcome: Elimination Half-Life Period (T1/2) of Bortezomib on Day 1 of Cycle 1
Description: The T1/2 is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal rate-constant (lambda[z]) of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Time Frame: 0 hour (Pre-dose) and 0.08, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours (post-dose) on Day 1 of Cycle 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Bortezomib
Number analyzed (Participants) | 10
Hours | 0.08 (0.07)

15. Primary Outcome: Elimination Half-Life Period (T1/2) of Bortezomib on Day 11 of Cycle 1
Description: as for outcome 14
Time Frame: 0 hour (Pre-dose) and 0.08, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours (post-dose) on Day 11 of Cycle 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Bortezomib
Number analyzed (Participants) | 10
Hours | 51.55 (87.20)

16. Primary Outcome: Terminal Rate Constant (Lambda[z]) of Bortezomib on Day 1 of Cycle 1
Description: Lambda(z) is defined as terminal rate-constant which reflect the speed of drug elimination in vivo (within the living), and is estimated by log-linear regression analysis of the terminal phase of the plasma concentration versus time curve for at least 3 points.
Time Frame: 0 hour (Pre-dose) and 0.08, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours (post-dose) on Day 1 of Cycle 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Per Hour
Arm/Group | Bortezomib
Number analyzed (Participants) | 10
Per Hour | 0.08 (0.07)

17. Primary Outcome: Terminal Rate Constant (Lambda[z]) of Bortezomib on Day 11 of Cycle 1
Description: as for outcome 16
Time Frame: 0 hour (Pre-dose) and 0.08, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours (post-dose) on Day 11 of Cycle 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Per Hour
Arm/Group | Bortezomib
Number analyzed (Participants) | 10
Per Hour | 0.01 (0.01)

18. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Time at Last Observed Quantifiable Concentration (AUC[0-t]) of Bortezomib on Day 1 of Cycle 1
Description: The AUC(0-t) is area under the plasma concentration-time curve from time zero to the last quantifiable concentration determined by the trapezoidal rule.
Time Frame: 0 hour (Pre-dose) and 0.08, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours (post-dose) on Day 1 of Cycle 1
Population: PP population included all the participants who received study medications as per the administration schedule and for whom blood samples were collected at all scheduled time points.
Measure: Mean (Standard Deviation); unit: Hour*ng per ml
Arm/Group | Bortezomib
Number analyzed (Participants) | 10
Hour*ng per ml | 51.86 (30.56)

19. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Time at Last Observed Quantifiable Concentration (AUC[0-t]) of Bortezomib on Day 11 of Cycle 1
Description: The AUC(0-t) is area under the plasma concentration-time curve from zero to the last quantifiable concentration determined by the trapezoidal rule.
Time Frame: 0 hour (Pre-dose) and 0.08, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours (post-dose) on Day 11 of Cycle 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Hour*ng per mL
Arm/Group | Bortezomib
Number analyzed (Participants) | 10
Hour*ng per mL | 190.39 (55.27)

20. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of Bortezomib on Day 1 of Cycle 1
Description: The AUC(0-infinity) is area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z), in which C(last) is the last observed quantifiable concentration.
Time Frame: Day 1 of Cycle 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Hour*ng per ml
Arm/Group | Bortezomib
Number analyzed (Participants) | 10
Hour*ng per ml | 106.99 (126.91)

21. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of Bortezomib on Day 11 of Cycle 1
Description: as for outcome 20
Time Frame: 0 hour (Pre-dose) and 0.08, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours (post-dose) on Day 11 of Cycle 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Hour*ng per ml
Arm/Group | Bortezomib
Number analyzed (Participants) | 10
Hour*ng per ml | 349.62 (178.81)

22. Primary Outcome: Area Under First Moment Plasma Concentration-Time Curve (AUMC) of Bortezomib on Day 1 of Cycle 1
Description: AUMC is defined as the area under first moment plasma concentration-time curve from time of dosing up to definite time t, to infinity, or to the time of last measurable concentration determined by the following equation: AUMC(0 to infinity)=Cntn/k elimination(el) + Cn/k(el^2) summation[(tn - tn^-1) (Cn^-1) (tn^-1)] + Cntn/2 where Cn=last quantifiable concentration, tn=time at which Cn is measured, k=rate constant.
Time Frame: 0 hour (Pre-dose) and 0.08, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours (post-dose) on Day 1 of Cycle 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Hour square*ng per ml
Arm/Group | Bortezomib
Number analyzed (Participants) | 10
Hour square*ng per ml | 20678.41 (54596.1)

23. Primary Outcome: Area Under First Moment Plasma Concentration-Time Curve (AUMC) of Bortezomib on Day 11 of Cycle 1
Description: as for outcome 22
Time Frame: 0 hour (Pre-dose) and 0.08, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours (post-dose) on Day 11 of Cycle 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Hour square*ng per ml
Arm/Group | Bortezomib
Number analyzed (Participants) | 10
Hour square*ng per ml | 39414.06 (51021.07)

24. Primary Outcome: Mean Residence Time (MRT) of Bortezomib in the Body on Day 1 of Cycle 1
Description: The MRT is the average time at which the number of absorbed molecules reside in the body, after single-dose administration, and calculated as AUMC(infinity)/AUC(infinity) where AUMC(infinity) is area under the plasma concentration-time first moment curve from time zero to infinite time and AUC(infinity) is the area under the plasma concentration-time curve from time zero to infinite time.
Time Frame: 0 hour (Pre-dose) and 0.08, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours (post-dose) on Day 1 of Cycle 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Bortezomib
Number analyzed (Participants) | 10
Hour | 65.97 (121.65)

25. Primary Outcome: Mean Residence Time (MRT) of Bortezomib in the Body on Day 11 of Cycle 1
Description: as for outcome 24
Time Frame: 0 hour (Pre-dose) and 0.08, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours (post-dose) on Day 11 of Cycle 1
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Bortezomib
Number analyzed (Participants) | 10
Hour | 88.74 (58.38)

26. Primary Outcome: Systemic Clearance (CL) of Bortezomib on Day 1 of Cycle 1
Description: Systemic CL is a quantitative measure of the rate at which a drug substance is removed from the body. The total systemic clearance after intravenous dose was estimated by dividing the total administered dose by the plasma AUC(0-infinity).
Time Frame: 0 hour (Pre-dose) and 0.08, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours (post-dose) on Day 1 of Cycle 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Liter per Hour
Arm/Group | Bortezomib
Number analyzed (Participants) | 10
Liter per Hour | 25.99 (18.54)

27. Primary Outcome: Systemic Clearance (CL) of Bortezomib on Day 11 of Cycle 1
Description: as for outcome 26
Time Frame: 0 hour (Pre-dose) and 0.08, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours (post-dose) on Day 11 of Cycle 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Liter per Hour
Arm/Group | Bortezomib
Number analyzed (Participants) | 10
Liter per Hour | 4.68 (2.46)

28. Primary Outcome: Volume of Distribution at Steady-State (Vss) of Bortezomib on Day 1 of Cycle 1
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state which is estimated by (D/AUC[0-infinity])*(AUMC[0-infinity])/AUC[0-infinity]) where D is the dose of study drug, AUMC(0-infinity) is the area under the first moment curve extrapolated to infinity and AUC(0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time.
Time Frame: 0 hour (Pre-dose) and 0.08, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours (post-dose) on Day 1 of Cycle 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Bortezomib
Number analyzed (Participants) | 10
Liter | 483.71 (403.04)

29. Primary Outcome: Volume of Distribution at Steady-State (Vss) of Bortezomib on Day 11 of Cycle 1
Description: as for outcome 28
Time Frame: 0 hour (Pre-dose) and 0.08, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours (post-dose) on Day 11 of Cycle 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Bortezomib
Number analyzed (Participants) | 10
Liter | 331.68 (85.81)

ADVERSE EVENTS:
Time Frame: Basleine up to Day 11 of Cycle 8
Arm/Group | Bortezomib
Serious Adverse Events (participants affected / at risk) | 14/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib (N=14)
Pancytopenia (Blood and lymphatic system disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 4
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Ammonia abnormal (Investigations) | 1
Blood albumin decreased (Investigations) | 1
Blood antidiuretic hormone abnormal (Investigations) | 1
Blood calcium increased (Investigations) | 1
Blood glucose decreased (Investigations) | 1
Blood potassium decreased (Investigations) | 2
Blood sodium increased (Investigations) | 2
Mini mental status examination abnormal (Investigations) | 1
Platelet count decreased (Investigations) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib (N=14)
Tachycardia (Cardiac disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 3
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 1
Gingival ulceration (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Oesophageal ulcer (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Chest pain (General disorders) | 4
Irritability (General disorders) | 1
Localised oedema (General disorders) | 2
Nodule (General disorders) | 1
Oedema (General disorders) | 2
Oedema peripheral (General disorders) | 4
Pain (General disorders) | 1
Pyrexia (General disorders) | 7
Device related infection (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 3
Infections - pathogen unspecified (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Salmonella bacteraemia (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 7
Blood albumin decreased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 1
Blood amylase increased (Investigations) | 1
Blood calcium decreased (Investigations) | 3
Blood calcium increased (Investigations) | 3
Blood cholesterol increased (Investigations) | 1
Blood creatinine abnormal (Investigations) | 1
Blood creatinine increased (Investigations) | 4
Blood glucose increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 1
Blood magnesium decreased (Investigations) | 1
Blood magnesium increased (Investigations) | 1
Blood phosphorus decreased (Investigations) | 2
Blood potassium decreased (Investigations) | 5
Blood sodium increased (Investigations) | 2
Blood triglycerides increased (Investigations) | 1
Blood uric acid increased (Investigations) | 3
Gamma-glutamyltransferase increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 9
Neutrophil count decreased (Investigations) | 11
Platelet count decreased (Investigations) | 10
Weight decreased (Investigations) | 4
White blood cell count decreased (Investigations) | 11
Anorexia (Metabolism and nutrition disorders) | 6
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 3
Hypoaesthesia (Nervous system disorders) | 6
Nervous system disorder (Nervous system disorders) | 5
Neuralgia (Nervous system disorders) | 7
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 3
Dysuria (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 3
Blood potassium increased (Investigations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less